CLINICAL TRIAL: NCT04012827
Title: A Single-arm, Open, Multicenter Study of Apatinib Mesylate Combined With Doxorubicin and Ifosfamide in Advanced Soft-tissue Sarcoma
Brief Title: Apatinib Mesylate Combined With Doxorubicin and Ifosfamide in Advanced Soft-tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xing Zhang, Vice director of department of medical sarcoma and melanoma,Principal Investigator,Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SunYat-senU-apatinib
Record Dates: First submitted 2019-07-07; First posted 2019-07-09 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — apatinib; Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib Mesylate Combined With Doxorubicin and Ifosfamide (Experimental): A course of treatment every 21 days. For patients with disease control (CR+ PR+SD) and tolerable adverse reactions after 6 courses of treatment, continuous drug use was considered by the researchers as inappropriate for patients to continue drug use or when the efficacy was assessed as disease progression (PD).No other antitumor treatment can be given during the treatment.
  Interventions: Drug: Apatinib Mesylate, doxorubicin, ifosfamide

INTERVENTIONS:
Drug: Apatinib Mesylate, doxorubicin, ifosfamide — Doxorubicin 50mg/m2 d1 , Ifosfamide 2.5g/m2 d1-3 , Apatinib mesylate 375mg qd
  Other Names: Apatinib

SUMMARY:
Apatinib mesylate is a multitarget receptor tyrosine kinase inhibitor. This trial is to evaluate the efficacy and safety of apatinib mesylate combined with doxorubicin and ifosfamide in the treatment of advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
Apatinib mesylate has demonstrated good efficacy and acceptable safety in patients with metastatic or recurrent soft tissue sarcoma (STS). A retrospective study has evaluated the efficacy of apatinib in the treatment of advanced soft tissue sarcoma. A total of 31 patients with soft tissue sarcoma were enrolled in this study, including 4 patients receiving apatinib first-line treatment, 8 patients receiving second-line treatment, and 19 patients receiving third-line or post-third-line treatment. The results showed that ORR 33.3%, DCR 75%, and mTTP 4.6 months (1.8-11.6 months). In another multicentric retrospective study of apatinib for osteosarcoma and soft tissue sarcoma, a total of 56 patients were enrolled and 44 were treated with apatinib monotherapy. The overall results showed that ORR was 62.5%, mPFS was 6.6 months, and mOS was 9.9 months. In a phase II multi-center single-arm study results published by Yang Jilong Yang et al at the 2018 AACR conference, ORR and DCR at 3 months also reached 13.95% and 81.39%, respectively. The end point assessment ORR was further increased to 15.25% at the end of the study, because some patients achieved partial remission after a long period of treatment, and the final DCR reached 57.63%. Apatinib had a significant effect in the treatment of stage IV osteosarcoma with failed chemotherapy. Jing Chen et al published a study researching the effectiveness and security in advanced sarcoma patients after apatinib treatment , the results show that 24.3% of subjects to achieve objective response, including 1 case of adenoid vesicular soft tissue sarcoma patients achieved CR, seven adenoid vesicular soft tissue sarcoma patients achieved the objective response, indicates that apatinib is effective and well tolerated in some specific sarcoma subtype.

In this study ,Apatinib mesylate combined with doxorubicin and ifosfamide regimens were evaluated in the treatment of advanced or inoperable STS to determine the potential to achieve better outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in this study and signed the informed consent;
2. The pathology diagnosed with at least one measurable lesion according to RECIST 1.1 standard. The pathology includes synovial sarcoma, leiomyosarcoma, angiosarcoma, undifferentiated pleomorphic sarcoma/malignant fibrous histiocytoma, liposarcoma, fibrosarcoma, clear cell sarcoma, epithelioid sarcoma, malignant peripheral nerve sheath tumor, undifferentiated sarcoma, rhabdomyosarcoma, dermatofibrosarcoma protuberans, ewing's sarcoma /primary neural ectoderm tumors, desmoplastic small round cell tumor, inflammatory myofibroblastic sarcoma, malignant solitary fibroma. Except for chondrosarcoma, osteosarcoma, malignant mesothelioma, alveolar soft tissue sarcoma, gastrointestinal stromal tumor;
3. Patients with recurrence after surgery or with lymph nodes or distant metastasis after imaging evaluation;
4. 18 ~ 70 years old; ECOG PS score: 0~1; Expected survival beyond 3 months;
5. Major organs functions should meet the following standards within 7 days before treatment:

(1) Blood routine examination standard (without blood transfusion within 14 days) : Hemoglobin (HB) ≥90g/L; The absolute value of neutrophils (ANC) ≥1.5×109/L; Platelet (PLT) ≥80 ×109/L.

(2) Biochemical examination shall meet the following standards: Total bilirubin (TBIL) ≤ 1.5 times ULN (Upper Limit Of Normal); alanine aminotransferase （ALT）and aspartate aminotransferase AST≤2.5 times ULN. If accompanied by liver metastasis, ALT and AST≤5 times ULN；Serum creatinine（Cr）≤1.5 times ULN or creatinine clearance rate (CCr)≥ 60ml/min；

(3) Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%).

6. Women of reproductive age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during and within 6 months after the study; Negative serum or urine pregnancy test within 7 days prior to study enrollment and must be non-lactating; Men should agree to use contraceptives during and within 6 months after the study period.

Exclusion Criteria:

1. Patients who have previously used apatinib mesylate;
2. Received any form of chemotherapy after recurrence or metastasis;
3. Patients previously treated with targeted drugs of vascular endothelial growth inhibitors, such as sunitinib, sorafenib, bevacizumab, imatinib, famitinib, pazopanib, regorafenib, and anlotinib.
4. Other malignancies that have occurred or are present at the same time within 5 years, except for cured cancers including carcinoma in situ of the cervix, non-melanoma skin cancer and superficial bladder tumor [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
5. Systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, and immunotherapy (or mitomycin C administration within 6 weeks before the treatment with the experimental drug), is planned within 4 weeks before enrollment or during the medication period of this study. In the first 4 weeks of enrollment, the patients were treated with field expanding radiotherapy (ef-rt) or the limited field radiotherapy designed to evaluate tumor lesions in the first 2 weeks of enrollment.
6. Accompanied by pleural effusion or ascites, causing respiratory syndrome (CTCAE grade 2 dyspnea [grade 2 dyspnea refers to shortness of breath when there is a small amount of activity; it affects instrumental daily life activities]);
7. Unrelieved toxic reactions caused by any previous treatment higher than CTCAE (4.1) level 1 or above, excluding hair loss;
8. Patients with multiple factors (such as inability to swallow, chronic diarrhea and intestinal obstruction) affecting oral drugs;
9. Patients with brain metastases with symptoms or with symptoms for less than 2 months;
10. Patients with any severe and/or uncontrolled disease, including:

1)Patients with unsatisfactory blood pressure control (systolic blood pressure 150 mmHg, diastolic blood pressure 100 mmHg);

2)Patients with grade I or above myocardial ischemia or myocardial infarction, arrhythmia (including QTC 480ms) and grade II congestive heart failure (NYHA classification);

3)Active or uncontrolled severe infection (CTCAE grade 2 infection);

4)Cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral treatment;

5) Renal failure requires hemodialysis or peritoneal dialysis;

6) Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;

7)Poor control of diabetes mellitus (FBG) > 10mmol/L);

8)Urine routine test indicated urine protein ++, and confirmed the 24-hour urine protein quantitative > 1.0g;

9)Patients with seizures requiring treatment;

11. Received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before enrollment;

12. Patients with any signs of bleeding constitution or medical history, regardless of the severity; Patients with any bleeding or bleeding event CTCAE level 3 within 4 weeks before enrollment have unhealed wounds, ulcers or fractures;

13. Hyperactive/venous thrombosis events within 6 months, such as cerebrovascular accidents (including temporary ischemic attack), deep venous thrombosis and pulmonary embolism;

14. Patients with active ulcer, intestinal perforation and intestinal obstruction;

15. Have a history of mental drug abuse and cannot quit or have mental disorder;

16. Participated in clinical trials of other anti-tumor drugs within 28 days before enrollment;

17.According to the judgment of the researcher, there are those who seriously endanger the safety of patients or affect the patients' completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 24 months
  Objective response rate is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.

SECONDARY OUTCOMES:
Progress free survival | From treatment until progression (up to 24 months)
  Progress free survival defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.
Overall Survival | From treatment until death (up to 24 months)
  Overall survival is defined as the time until death due to any cause.
Disease Control Rate | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China